CLINICAL TRIAL: NCT03993600
Title: MucoSWEATomics New Markers of CFTR Function in Sweat: Value for Diagnosis and Efficacy of Target Therapies
Brief Title: New Markers of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Function in Sweat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Université de Liège (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/09OCT/374
Record Dates: First submitted 2019-05-14; First posted 2019-06-20 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis; Biomarkers
Keywords: cystic fibrosis; sweat; sweat glands; omics analysis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Three groups will be done : healthy volunteer, cystic fibrosis patient and heterozygotes subject
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Sham Comparator): sweat test and skin biopsy
  Interventions: Diagnostic Test: Sweat test (Macroduct Sweat Collection System) and skin biopsy (Punch Biopsy)
- Patients with Cystic fibrosis (Experimental): sweat test and skin biopsy
  Interventions: Diagnostic Test: Sweat test (Macroduct Sweat Collection System) and skin biopsy (Punch Biopsy)
- Heterozygotes subjects (Experimental): sweat test and skin biopsy
  Interventions: Diagnostic Test: Sweat test (Macroduct Sweat Collection System) and skin biopsy (Punch Biopsy)

INTERVENTIONS:
Diagnostic Test: Sweat test (Macroduct Sweat Collection System) and skin biopsy (Punch Biopsy) — three groups:
  1. Healthy volunteers
  2. Patients with Cystic fibrosis
  3. Heterozygous subjects

SUMMARY:
The aim of the study is to identify new biomarkers of CFTR function in sweat and in sweat gland.

DETAILED DESCRIPTION:
Sweat is a watery solution containing trace amounts of proteins and peptides that may contribute to the antimicrobial defense system of the skin barrier, playing a role in innate immune responses against potential pathogens. The peptide and metabolite composition of sweat has not been fully explored. Evidence suggests that the composition of the skin barrier could vary with diseases. The causes and consequences of the changes of sweat proteins and peptides in humans are unknown. This clinical trial will focus on multiomics analysis of sweat, mainly of the antimicrobial peptides that play a key role in the host-pathogen interaction. Antioxidants, anti-bacterial and anti-inflammatory compounds may contribute to the regulation of systemic inflammation and pathophysiological disorders. In cystic fibrosis, inflammatory responses are altered, exaggerated and persistent, even in the absence of infection. It is therefore relevant to study the influence of CFTR mutations on the profile of antimicrobial peptides expressed in sweat. The clinical study will potentially lead to the discovery of novel non-invasive biomarkers of the disease in sweat.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged of 18 years or more.
* The patients with cystic fibrosis must have a confirmed diagnosis, be clinically stable, have a Forced Expiratory Volume in one second (FEV1) ≥ 30 and an O2 saturation ≥ 92%. F508del homozygous will been tested.
* Heterozygosity (parents of patients) will be confirmed by the presence of a single F508del mutation.

Exclusion Criteria:

* Presence of an acute infection
* Pregnancy and lactation
* Subjects currently included in another clinical trial
* Subjects with forearm skin alterations
* Subjects with signs of dehydration
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistical analysis | one day
  The assessment of the quantity of sweat secreted will be measured in mg with a scale, the sweat chloride concentration will be done by coulometric titration and expressed in mmol/L.

SECONDARY OUTCOMES:
Proteomics, peptidomics and metabolomics analysis on sweat and sweat glands | 2 years
  The quantity of total protein will be analysed with a colorimetric assay and will be expressed in mg/ml.
  The identification of the different protein will be performed with different software, databases and algorithms such as Proteome Discoverer (version 1.4.1.14), Mascot software (version 2.2.0.6), MaxQuant (version 1.5.2.8), Andromeda, Uniprot, LFQ and Perseus (version 1.5.0.15).

CONTACTS AND LOCATIONS:
Overall Officials: Teresinha Leal, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No